CLINICAL TRIAL: NCT04114890
Title: The Pharmacokinetic Parameters of Tenofovir (TFV) in Maternal Blood and Breast Milk in Women Treated With Daily Tenofovir Disoproxil Fumarate (TDF; 300mg) for Prevention of Mother to Child Transmission (PMTCT) of Hepatitis B Virus (HBV) Mono-infection
Brief Title: Tenofovir in Pregnancy to Prevent Mother to Child Transmission of Hepatitis B.
Acronym: PK-TDF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VIR19001
Record Dates: First submitted 2019-09-18; First posted 2019-10-03 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis B; Tenofovir; Pregnancy
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant woman with second trimester and third trimester (Experimental)
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate 300 mg once daily and will continue until one month after delivery

SUMMARY:
Hepatitis B virus (HBV) can be asymptomatic for years but can also lead to chronic hepatitis, hepatocellular carcinoma, and liver failure and death and cannot be eradicated with the current therapy. Chronic maternal HBV infection is an important source of perinatal transmission in regions of high HBV prevalence. In antenatal clinics at Shoklo Malaria Research Unit (SMRU), the Hepatitis B (HB) surface antigen (sAg) prevalence is 8.3% with a HB e-antigen (HBeAg) prevalence of 32.7% in those positive for HBsAg in 2012-2014. Perinatal infection occurs in 70-90% of women with HBeAg positive chronic HBV compared with 0-30% in those with HBeAg negative chronic HBV (inactive carriers). These infection rates reflect, in part, the failure of maternal and child health programs to prevent perinatal transmission with hepatitis B immunoglobulin (HBIG) and HB vaccines. Prevention of mother to child transmission (PMTCT) fails in an estimated 8-32% of cases with adequate preventive techniques. Antiretrovirals, like tenofovir (TFV) that is administered as the prodrug Tenofovir Disoproxil Fumarate (TDF), are active against HBV and may reduce the risk of HBV transmission at birth if offered at the right time in pregnancy.

One of the major gaps in implementing this strategy is adequate pharmacokinetic (PK) data in pregnant women that informs correct dosing. One recently published population PK study in 154 women who provided maternal blood samples (32 and 36 weeks of pregnancy, at delivery, and at 1 and 2 months post-partum) reported a tenofovir area under curve (AUC) 0-24 that was estimated to be 20% (95% CI, 19-21%) lower during pregnancy than during post-partum suggesting no dose adjustments are needed in 3rd trimester. Most PK studies for TDF in pregnancy have been for Human Immunodeficiency Virus type 1 (HIV-1) infections. However, these patients often receive additional antiretroviral medications, preventing conclusions on PK parameters of Tenofovir (TFV) alone. Doses that are optimal for HIV may not be appropriate for HBV.

When TDF is administered during pregnancy and potentially during lactation, it is important to establish the infant drug exposure. Previous human studies have shown that antiretrovirals administered to lactating mothers are present in the breast milk and have detected a low TDF breast milk concentration representing 0.03% or less of the proposed infant dosage. However, there is no data on this subject in therapeutic treatment of HBV infected women. In resource poor settings TDF administration will be ceased after 1 month post-partum. While there is some understanding of what happens to viral load post cessation in non-pregnant individuals, post-partum TDF cessation is less well understood and may be affected by differences in immunity. With breastmilk as the primary source of nutrition for babies in resource limited settings, it is important to know the viral exposure from breastmilk, if any, as these settings may also have problems achieving birth dose, HBIG and completion of the recommended three doses of vaccine.

The investigators propose a dense PK study of once daily TDF 300 mg during pregnancy given for PMTCT of HBV mono-infection. Tenofovir PK will be measured in maternal blood samples in steady-state, in the 2nd and 3rd trimesters and post-partum. The presence of HBV DNA in blood and breast milk will also be explored in women after cessation of treatment until 6 months post-partum.

DETAILED DESCRIPTION:
Participants with HBV mono infection and a measurable HBV DNA viral load attending SMRU antenatal clinics (ANC) on the Myanmar-Thailand border will be invited if they have a gestational age of at least 20 weeks. A total of 24 women: 12 participants enrolled in 2nd trimester (EGA 20-<24 weeks) and 12 enrolled in 3rd trimester (EGA 28-<36) with complete samples are required.

Women, identified by routine antenatal care screening for HBV will be invited to participate if they are HBsAg positive and meet the inclusion and exclusion criteria. Participants will be provided TDF 300mg daily and will continue TDF treatment until one month after delivery. The TFV concentrations will be measured monthly before delivery, at delivery, in cord blood and 1 and 2 months postpartum. Additional dense PK blood sampling will be done in the second and third trimester and postpartum. Breast milk samples timed with mother blood and infant blood samples will be included to measure drug concentrations in breastmilk as possible presence of HBV DNA viral in breastmilk following cessation of TDF.

The dense sampling for pharmacokinetics assessments will occur at least after 2 weeks of TDF treatment in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks postpartum. The dense sampling will entail twelve blood samples in a 24 hour period (24ml of blood in total). Women will be counseled about the importance of adherence. Direct Observed Treatment (DOT) in the 3 days prior to the dense blood sampling will be performed. The woman can choose to be admitted for these days or if a home visitor lives close enough be supervised at home.

The follow-up for women will be until 6 months post-partum, to check for flares. TFV concentrations will be collected by venous blood testing but an indwelling catheter can be used during the rich sampling 24 hour period. Infants will be followed up from delivery, and at 1, 2, 4 and 6 months of age for vaccination and growth. Infant drug exposure is measured at month 1 and HBV DNA will be measured at birth from cord blood and HBsAg by venepuncture at 2 months of age.

Funder & grant reference number: iTPA Award (grant ref. no. WT-iTP-2019/006)

ELIGIBILITY:
Inclusion Criteria:

* Single viable pregnancy at enrollment day
* Estimated Gestational Age (EGA) 20-<24 weeks for 2nd trimester or EGA 28-<34 for 3rd trimester
* Willing and able to give informed consent for participation in the study
* Hepatitis B infected (HBsAg and HBeAg confirmed positive or HBsAg confirmed positive and HBV DNA detected in HBeAg negative)
* Burmese and Karen female, 16-49 years (inclusive)
* Willing to take TDF daily during pregnancy
* Plans to deliver at SMRU clinics

Exclusion Criteria:

* Undetectable HBV DNA in HBeAg negative women
* HIV infected or other chronic illness incompatible with the study requirements or receiving Immunosuppressive therapy
* Creatinine at screening >1 mg/dL
* Serum phosphate <2.4 mg/dL
* History of chronic kidney disease

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve [AUC] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.
Maximum (peak) plasma drug concentration [Cmax] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.
Minimum plasma drug concentration [Cmin] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.
Initial (fictive) or back-extrapolated plasma drug concentration at time zero [C0] | At pre-dose (in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.)
Plasma drug concentration at time 24 [C24] | At 24 hours post-dose (in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.)
Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]) [Cthrough] | At the end of a dosing interval at steady state
Apparent total clearance of the drug from plasma after oral administration [CL/F] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.
Elimination half-life [t½] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.
Time to reach maximum (peak) plasma concentration following drug administration [tmax] | At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose in second trimester between 22-26 weeks gestation, in third trimester between 30-38 weeks gestation, and 4 weeks post-partum.

SECONDARY OUTCOMES:
Maternal breastmilk TFV concentrations | 1 month post-partum
Milk to maternal plasma concentration ratios (M/P) | 1 month post-partum
Infant plasma drug concentration | At 1 month of life
HBV DNA in blood and breastmilk | At delivery and 1, 2, 3, 4, 5, and 6 months post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research unit (SMRU) clinics, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Subject's clinical data and results from blood analyses stored in our database may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the subject.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04114890/Prot_SAP_001.pdf